CLINICAL TRIAL: NCT00718640
Title: Safety and Efficacy of Velcade in Relapsed and/or Refractory Multiple Myeloma Patients With Impaired Renal Function
Brief Title: An Efficacy and Safety Study of Bortezomib in Participants Previously Treated for Multiple Myeloma With Limited Kidney Function
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study stopped due to lagging enrolment.
Sponsor: Janssen-Ortho Inc., Canada (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR015082; 26866138MMY2052
Record Dates: First submitted 2008-07-17; First posted 2008-07-21 (Estimated); Results first posted 2013-08-28 (Estimated); Last update posted 2013-10-29 (Estimated); Status verified 2013-09

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; Velcade; Bortezomib; Dexamethasone
MeSH Terms: conditions — Multiple Myeloma | interventions — Dexamethasone; Bortezomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Bortezomib and Dexamethasone (Experimental): Bortezomib 1.3 milligram (mg) per meter^2 (m^2) bolus (a large amount) intravenous (into the vein) injection will be administered once daily on Days 1, 4, 8 and 11 of each 21-day cycle with addition of Dexamethasone 20 mg per day administered orally, once daily on Days 1 and 2, Days 4 and 5, Days 8 and 9 and Days 11 and 12 of each 21-day cycle as per Investigator's discretion for those participants who experience disease progression after treatment completion up to Cycle 2 or have no change from Baseline after completion of at least 4 cycles. The treatment will be given up to 8 cycles (24 weeks).
  Interventions: Drug: Dexamethasone; Drug: Bortezomib

INTERVENTIONS:
Drug: Dexamethasone — Dexamethasone 20 mg per day will be administered orally on Days 1 and 2, Days 4 and 5, Days 8 and 9 and Days 11 and 12 of each 21-days cycle as per Investigator's discretion for those participants who experience disease progression after treatment completion up to Cycle 2 or have no change from Baseline after completion of at least 4 cycles. The treatment will be given up to 8 cycles (24 weeks).
Drug: Bortezomib — Bortezomib 1.3 milligram per meter^2 (mg/m^2), bolus intravenous injection will be administered on Days 1, 4, 8 and 11 of each 21-day cycle and up to 8 cycles.
  Other Names: Velcade

SUMMARY:
The purpose of this study is to evaluate the effectiveness and safety of bortezomib in participants previously treated for multiple myeloma (cancer of plasma cells in bone marrow causing numerous tumors and characterized by the presence of abnormal proteins in the blood) with limited kidney function.

DETAILED DESCRIPTION:
This is an open label (all people know the identity of the intervention), multi-center (study conducted at multiple sites), non-comparative, single arm study of bortezomib. The study consists of 3 phases: Screening phase (21 days before Day 1 of cycle 1); Treatment phase (consist of 8 cycles each cycle of 21 days or until disease progression or unacceptable toxicity); and a Follow-up phase (for participants with positive treatment response or stable disease at the final visit). Follow-up for disease progression will be done in every 3 months up to 2 years. Participants who will experience disease progression after completing at least 2 cycles of bortezomib treatment or have no change from baseline in stable disease after completing at least 4 cycles or as per Investigator's discretion will receive dexamethasone. Efficacy will be primarily evaluated by percentage of participants with renal compromised Multiple Myeloma by International Myeloma Working Group (IMWG) uniform response criteria. Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Participants diagnosed with symptomatic multiple myeloma based on the International Myeloma Working Group (IMWG) criteria; greater than or equal to 10 percent plasma cells in the bone marrow (or tissue biopsy) detected, monoclonal protein in the serum or urine and the, presence of end-organ injury
* Participants with measurable disease defined by at least 1 of the following 5 measurements: a) serum M-protein greater than or equal to 1 gram per deciliter (g/dl), b) Urine M Protein greater than or equal to 200 milligram per 24 hour, c) Serum free light chain (FLC) assay: Involved FLC level greater than 10 mg per dl (mg/dl) provided serum FLC ratio is abnormal, d) Bone marrow plasma cells greater than or equal to 30 percent
* Participants who received at least 1 prior line of chemotherapy for multiple myeloma and, is refractory to or has relapsed after the last therapy
* Participants with Karnofsky performance status greater than 60 or Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
* Participants with calculated or measured creatinine clearance of less than or equal to 30 mililiter per minute (ml/min). During the screening period, 2 measures of creatinine clearance at least 7 days apart must be obtained, and both must be less than 30 ml/min

Exclusion Criteria:

* Participants who had received bortezomib in previous clinical trial and best response was progressive disease or experienced one or more serious events
* Participants who received nitorsoureas within 6 weeks, or 2 consecutive weeks of intense corticosteroids, or immunotherapy or antibody therapy within 4 weeks before enrolment
* Participants with history of allergic reaction attributable to compounds containing boron or mannitol
* Participants with peripheral neuropathy of Grade 2 or greater intensity at the time of signing informed consent form
* Pregnant or breast-feeding female participants

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2007-10; Primary Completion 2009-12 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Inc. Clinical Trial, Study Director — Janssen Inc.
Locations (5):
- Canada (5):
  - New Westminster, British Columbia
  - Vancouver, British Columbia
  - London, Ontario
  - Greenfield Park, Quebec
  - Saint John

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Bortezomib and Dexamethasone
Started | 10
Completed | 3
Not Completed | 7
Not completed — Adverse Event | 4
Not completed — Death | 1
Not completed — Unresolved toxicity after 2 weeks | 2

BASELINE CHARACTERISTICS:
Arm/Group | Bortezomib and Dexamethasone
Number analyzed (Participants) | 10
Age, Customized [Number; unit: participants]
  < 65 | 1
  Between 65-69 | 1
  Between 70-74 | 4
  >=75 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 4

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Renal Compromised Multiple Myeloma by International Myeloma Working Group (IMWG) Uniform Response Criteria
Description: The IMWG uniform response criteria define; Complete response(CR) as negative immunofixation on serum and urine, disappearance of any soft tissue plasmacytomas and <5% plasma cells in bone marrow(BM). Stringent CR as CR+normal free light chain ratio and absence of clonal cells in BM Very good partial response (PR) as serum and urine M-protein (monoclonal paraprotein) detectable by immunofixation but not on electrophoresis or 90% or >reduction in serum and urine M-protein level <100 milligram(mg) per 24 hour(hr).PR as <=50% reduction of serum and <= 90% of urine M-protein or up to <200 mg/24 hr.
Time Frame: Week 24 or Early termination visit (30-45 days after last dose)
Population: The study was terminated. Due to insufficient number of participants, the outcome measure data was not analyzed.
Arm/Group | Bortezomib and Dexamethasone
Number analyzed (Participants) | 0

2. Secondary Outcome: Best Response to Treatment
Description: It was assessed by IMWG criteria. It defines complete response as negative immunofixation on the serum and urine and disappearance of any soft tissue plasmacytomas and <5% plasma cells in bone marrow. Very good partial response as serum and urine M-protein detectable by immunofixation but not on electrophoresis or 90% or > reduction in serum and urine M-protein level<100 mg per 24 hour. Partial Response as <=50% reduction of serum M-protein and reduction in 24-hour urinary M-protein by <=90% or to <200mg per 24 hr.
Time Frame: Day 1 of Cycle 1, 2, 3, 4, 5, 5, 6, 7, 8 and Final/Early termination visit (30-45 days after last dose)
Population: The study was terminated. Due to insufficient number of participants, the outcome measure data was not analyzed.
Arm/Group | Bortezomib and Dexamethasone
Number analyzed (Participants) | 0

3. Secondary Outcome: Time to Progression (TTP) of Disease
Description: The TTP was defined as the time from the date of starting treatment until the date of first documented evidence of progression of disease or death.
Time Frame: Day 1 (Start of treatment) until the date of first documented evidence of progression of disease or death
Population: The study was terminated. Due to insufficient number of participants, the outcome measure data was not analyzed.
Arm/Group | Bortezomib and Dexamethasone
Number analyzed (Participants) | 0

4. Secondary Outcome: Duration of Response
Description: The duration of Response was defined as the time of first recorded achievement of a particular response level, which was defined according to IMWG uniform response criteria, as either complete response, stringent complete response, very good partial response or partial response included only responding participants, until the participants were assessed to have progressive disease.
Time Frame: Day 1 (Start of treatment) until the date of first documented achievement of response
Population: The study was terminated. Due to insufficient number of participants, the outcome measure data was not analyzed.
Arm/Group | Bortezomib and Dexamethasone
Number analyzed (Participants) | 0

5. Secondary Outcome: Eastern Cooperative Oncology Group Performance Status (ECOG PS) Score
Description: The ECOG PS Score 0 versus 1, wherein 0 signifies fully active, able to carry all pre-disease performance without restriction and 1 signifies restriction in physically strenuous activity but ambulatory (able to walk) and able to carry out work on a light or sedentary nature.
Time Frame: Day 1 of Cycle 1, 3, 5, 7 and Final visit/Early termination visit (30-45 days after last dose)
Population: The study was terminated. Due to insufficient number of participants, the outcome measure data was not analyzed.
Arm/Group | Bortezomib and Dexamethasone
Number analyzed (Participants) | 0

6. Secondary Outcome: Karnofsky Performance Status (KPS) Score
Description: The KPS is used to quantify participant's general well-being and activities of daily life and participants are classified based on their functional impairment. KPS score is 11-level score which ranges between 0 (death) to 100 (no evidence of disease). Higher score means higher ability to perform daily tasks.
Time Frame: Day 1 of Cycle 1, 3, 5, 7 and Final visit (30-45 days after last dose) or early termination visit
Population: The study was terminated. Due to insufficient number of participants, the outcome measure data was not analyzed.
Arm/Group | Bortezomib and Dexamethasone
Number analyzed (Participants) | 0

7. Secondary Outcome: Quality of Life Assessment by QLQ C-30
Description: The quality of life was assessed by the questionnaire QLQ C-30 designed by European Organization for the Research and Treatment of Cancer (EORTC). The EORTC QLQ-C30 is a 30-item questionnaire to assess the overall quality of life in cancer participants. Most questions used 4-point scale (1 'Not at All' to 4 'Very Much'); 2 questions used 7-point scale (1 'Very Poor' to 7 'Excellent'). Scores are averaged, and transformed to 0-100 scale; higher score for a symptom scale like the fatigue scale is equal to higher level of symptomatology or problems.
Time Frame: Final Visit/Early termination visit (30-45 days after last dose)
Population: The study was terminated. Due to insufficient number of participants, the outcome measure data was not analyzed.
Arm/Group | Bortezomib and Dexamethasone
Number analyzed (Participants) | 0

8. Secondary Outcome: Quality of Life Assessed by Euro Quality of Life (EQ-5D)
Description: The EQ-5D is a participant rated questionnaire to assess health-related quality of life in terms of a single utility score. It assesses level of current health for 5 domains: mobility, self-care, usual activities, pain and discomfort, and anxiety and depression where 1=better health state (no problems), 3=worst health state. Scoring formula was developed by Euro quality of life group which assigns a utility value for each domain in profile. Score is transformed and results in a total score range -0.594 to 1.000; higher score indicates a better health state.
Time Frame: Quality of Life (EQ-5D) Final Visit/Early termination visit (30-45 days after last dose)
Population: The study was terminated. Due to insufficient number of participants, the outcome measure data was not analyzed.
Arm/Group | Bortezomib and Dexamethasone
Number analyzed (Participants) | 0

9. Secondary Outcome: Renal Function
Description: Renal function was analysed by creatinine clearance. Creatinine clearance was calculated by Cockroft-Gault fourmula. Creatinine clearance is equal to 140 minus age multiplied by weight and constant (1 for men and 0.85 for women) divided by creatinine in (micro mole per liter)
Time Frame: Day 1 of Cycle 1, 2, 3, 4, 5, 5, 6, 7, 8 and Final/Early termination visit (30-45 days after last dose)
Population: The study was terminated. Due to insufficient number of participants, the outcome measure data was not analyzed.
Arm/Group | Bortezomib and Dexamethasone
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Day 1 up to 30 days after last dose of study medication
Arm/Group | Bortezomib and Dexamethasone
Serious Adverse Events (participants affected / at risk) | 4/10
Other Adverse Events (participants affected / at risk) | 9/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bortezomib and Dexamethasone (N=10)
Pneumonia (Infections and infestations) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Renal impairment (Renal and urinary disorders) | 1
Hypertension (Vascular disorders) | 1
Muscle weakness (Musculoskeletal and connective tissue disorders) | 1
Depressed level of consciousness (Nervous system disorders) | 1
Aphasia (Nervous system disorders) | 1
Speech disorder (Nervous system disorders) | 1
Confusion state (Psychiatric disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bortezomib and Dexamethasone (N=10)
Hypotension (Vascular disorders) | 1
Orthostatic hypotension (Vascular disorders) | 1
Hypertension (Vascular disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Mood altered (Psychiatric disorders) | 1
Confusional state (Psychiatric disorders) | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1
Neuropathy peripheral (Nervous system disorders) | 1
Neuralgia (Nervous system disorders) | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2
Hypokalaemia (Metabolism and nutrition disorders) | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 1
Anorexia (Metabolism and nutrition disorders) | 1
International normalised ratio increased (Investigations) | 1
Blood creatinine increased (Investigations) | 4
Blood albumin decreased (Investigations) | 1
Contusion (Injury, poisoning and procedural complications) | 1
Herpes zoster (Infections and infestations) | 1
Bacteraemia (Infections and infestations) | 1
Fatigue (General disorders) | 2
Asthenia (General disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 3
Lymphopenia (Blood and lymphatic system disorders) | 1
Leukopenia (Blood and lymphatic system disorders) | 1
Anaemia (Blood and lymphatic system disorders) | 2

LIMITATIONS AND CAVEATS:
Participants' recruitment was limited due to pre-defined criteria of renal disease and requirement of repeated evaluation of creatinine clearance. Due to insufficient number of participants the outcome measure data was not analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No